CLINICAL TRIAL: NCT01883869
Title: XANTHIPPE: Examining the Effect of Ticagrelor on Platelet Activation, Platelet-Leukocyte Aggregates, and Acute Lung Injury in Pneumonia
Brief Title: Targeting Platelet-Leukocyte Aggregates in Pneumonia With Ticagrelor
Acronym: XANTHIPPE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Susan Smyth, Principle Investigator, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-0374-F6A
Record Dates: First submitted 2013-05-01; First posted 2013-06-21 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Pneumonia; Community Acquired Pneumonia; Hospital Acquired Pneumonia; Acute Lung Injury
Keywords: Platelet inhibition; Platelet-leukocyte aggregates; Platelet-neutrophil aggregates; CAP; HAP; ALI; Blood Platelets
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia; Healthcare-Associated Pneumonia; Acute Lung Injury | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ticagrelor (Experimental): 180 mg orally once and then 90 mg orally daily for 7 days or until hospital discharge if sooner
  Interventions: Drug: ticagrelor
- placebo (Placebo Comparator): One loading dose and then daily for 7 days or until hospital discharge if sooner
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ticagrelor
  Other Names: Brilinta
  Arms: ticagrelor
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
The hypothesis to be tested is that ticagrelor (Brilinta™) will reduce platelet activation and markers of inflammation in patients with pneumonia.

DETAILED DESCRIPTION:
While it is well established that platelets are integral to hemostasis, more recent evidence points to an important role for platelets in inflammation and immunity. Platelet activation and sequestration in pulmonary tissue is a key feature in inflammatory or infectious states such as sepsis and acute respiratory distress syndrome (ARDS). Platelets may mediate acute lung injury (ALI) by recruiting neutrophils, triggering neutrophil extracellular DNA nets, and releasing granule contents and microparticles. Anti-platelet therapy in this setting may prevent platelet activation, platelet - leukocyte aggregate formation, and inflammation.

The objective of this pilot study is to determine if ticagrelor therapy in individuals with pneumonia reduces markers of platelet activation, platelet-leukocyte aggregates, inflammation, acute lung injury, and lung mechanics. Because the benefit of anti-platelet therapy may the greatest in patients with more significant lung injury, the investigators will enroll patients with community-acquired pneumonia (CAP) requiring hospitalization or patients with hospital acquired pneumonia (HAP) within 48 hours of diagnosis. On study day 1, subjects will be randomized to receive ticagrelor (180 mg load and 90 mg BID) or placebo. Study medication (ticagrelor or placebo) will be administered twice daily on days 2 - 7 or until hospital discharge, if sooner than 7 days. Blood will be collected and assays performed on day 1 prior to study medication administration (baseline), day 2, 3, 7, day of discharge (if before 7 days), and 30 days for analysis of platelet count, markers of platelet activation, platelet - leukocyte interactions, biomarkers of inflammation, and measurements of lung mechanics.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older
* Subjects must diagnosed with Community acquired pneumonia (CAP) or hospital acquired pneumonia (HAP) within 48 hours of diagnosis or presentation to hospital.
* Pneumonia will be defined as patients with a new radiographic finding(s) consistent with pneumonia and at least two of the following signs.

  1. Cough
  2. Fever: axillary temperature >37.5ºC or tympanic temperature >38.5ºC
  3. Hypothermia: axillary temperature <34ºC or tympanic temperature <35ºC.
  4. Purulent sputum production or respiratory secretion.
  5. Total peripheral white blood cell (WBC) count >10,000/mm3; or >15% band forms, regardless of total peripheral white count; or leucopenia with total WBC < 4500/mm
  6. Auscultatory findings on pulmonary examination of rales and/or evidence of pulmonary consolidation (dullness on percussion, bronchial breath sounds, or egophony)
  7. Hypoxemia - defined as partial O2 pressure <60mmHg while the patient was breathing normal air or a decrease in the partial O2 pressure of >= 25% from an initial range.

Exclusion Criteria:

1. Contraindication to ticagrelor (hypersensitivity or reaction to ticagrelor or another P2Y12 antagonist)
2. Active bleeding or major bleeding history (e.g. intracranial bleeding)
3. Clinically important anemia or thrombocytopenia (platelet count <30)
4. Surgery within 30 days or anticipated major surgery (Thoracic, Abdominal, Brain; placement of lines, tracheostomy, and chest tubes are not considered major).
5. Oral anticoagulant therapy that cannot be stopped.
6. Inability or unwillingness of treating physician to reduce dose of aspirin to 81mg.
7. Fibrinolytic therapy in the last 24 hours.
8. Increased risk of bradycardic events - 2nd or 3rd degree heart block, bradycardia induced syncope - unless pacemaker in place.
9. Underlying immunodeficiency (HIV, neutropenia, receiving immunomodulating agents, active hematologic malignancy, functional or anatomical asplenia and hypogammaglobulinemia).
10. Moderate or severe liver disease defined by Child Pugh score >7 using data from outpatient setting or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 fold upper limits of normal.
11. Renal dialysis
12. Concomitant therapy with strong CYP3A inhibitors; ketoconazole, itraconazole, voriconazole, saquinavir, nelfinavir, indinavir, or atazanavir.
13. Concomitant therapy with CYP3A substate with narrow therapeutic window: cyclosporin, quinidine.
14. Concomitant therapy with CYP3A inducer; rifampin/rifampicin, phenytoin, carbamazepine.
15. Pregnancy or lactation
16. Active treatment for cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Platelet-Leukocyte Aggregates | 30 day
  Platelet-leukocyte aggregates will be measured by flow cytometry.

SECONDARY OUTCOMES:
Platelet function tests | 30 day
  Platelet function will be monitored by aggregation and by measuring markers of platelet secretion
Systemic inflammation | 30 day
  Markers of inflammation will be measured in plasma or serum
Lung function | During hospital stay up to 30 days.
  In non-ventilated patients, spirometry, maximal voluntary ventilation, maximal inspiratory and expiratory pressure generation, and P/F ratio (PaO2/FiO2)
  In ventilated patients, respiratory system static compliance, airway resistance, oxygenation index (PaO2/FiO2), and maximal inspiratory and expiratory pressure generation.

OTHER OUTCOMES:
Significant Bleeding Event | 30 days
  The PLATO definition of bleeding will be used to classify events. Life-threatening bleeding is defined as fatal or intracranial or intrapericardial with cardiac tamponade or hypovolemic shock, or severe hypotension requiring pressors or surgery, decrease in hemoglobin of >50mg/ml or transfusion of ≥ 4units of packed red blood cells(pRBCs).
  Major bleeding is defined as significantly disabling (intraocular with permanent vision loss), 30 - 50 mg/ml decrease in hemoglobin, or transfusion of 2 - 3 U pRBCs.
  Minor bleeding will be captured using PLATO bleeding definition of bleeding that requires medication intervention to stop or treat.
Mechanical Ventilation | 30 days
  mechanical ventilation or ventilator free days at day 30
Sepsis | 30 days
  Diagnosis of Sepsis
Mortality | 30 days
Major Cardiovascular Event | 30 days
  Major cardiovascular event can by myocardial infarction, stroke, or life threatening arrhythmia.

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Smyth, MD PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky Hospitals, Lexington, Kentucky
  - University of Kentucky Hospital, Lexington, Kentucky

REFERENCES:
- [Derived] Sexton TR, Zhang G, Macaulay TE, Callahan LA, Charnigo R, Vsevolozhskaya OA, Li Z, Smyth S. Ticagrelor Reduces Thromboinflammatory Markers in Patients With Pneumonia. JACC Basic Transl Sci. 2018 Aug 28;3(4):435-449. doi: 10.1016/j.jacbts.2018.05.005. eCollection 2018 Aug. PMID 30175268